CLINICAL TRIAL: NCT01653847
Title: Impact of Two Prednisone-free Maintenance Immunosuppressive Regimens With Reduced Dose FK506+Everolimus vs. Standard Dose Tacrolimus (FK506)+ Mycophenolate Mofetil (MMF) on Subpopulation of T and B Cells, Renal Allograft Function and Gene Expression Profiles in Renal Allograft Biopsies at 12 Months Post-transplant. Prospective Single Center Study in Recipients of Renal Transplant Allograft.
Brief Title: Study in Recipients of Renal Transplant Allograft to Evaluate the Impact of Two Immunosuppressive Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Lorenzo Gallon, Associated Professor of Transplant Nephrology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Novartis- Everolimus
Record Dates: First submitted 2012-04-04; First posted 2012-07-31 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: End Stage Renal Failure With Renal Transplant
Keywords: transplant; kidney; renal disease
MeSH Terms: conditions — Kidney Diseases | interventions — Tacrolimus; Mycophenolic Acid; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Tacrolimus with MMF. (Active Comparator): This group will receive a standard dose Tacrolimus and MMF. This will follow standard of care protocol at Northwestern Memorial Hospital's Comprehensive Transplant Center.
  Interventions: Drug: Tacrolimus with MMF
- Group 2: Tacrolimus with Everolimus (Active Comparator): This group will receive a low dose Tacrolimus with concentration controlled Everolimus
  Interventions: Drug: Group 2: Tacrolimus with Everolimus.
- Donors (No Intervention): One time blood samples will be collected from kidney donors to recipients in this study

INTERVENTIONS:
Drug: Tacrolimus with MMF — Standard dose Tacrolimus and MMF. This will follow standard of care procedures at Northwestern Memorial Hospital's Comprehensive Transplant Center. MMF trough or area under the concentration time curve (AUC) shall not be used to adjust dosing. In this group, Tacrolimus will be initiated according to our practice. The Tacrolimus dose will be adjusted from day 3 on to achieve a target whole blood trough concentration of 8 ng/mL to 10 ng/mL. From month 2 until Month 6, the target Tacrolimus trough level will be reduced to 6 ng/mL to 8 ng/mL. After month 6, the target level of Tacrolimus will be reduced to 4 ng/mL to 8 ng/mL.
  Other Names: Tacrolimus; FK 506; mycophenolate mofetil; MMF
  Arms: Group 1: Tacrolimus with MMF.
Drug: Group 2: Tacrolimus with Everolimus. — From day 5 on, the starting dose of Everolimus (0.75 mg bid) will be increased if the trough level is < 3 ng/mL, or reduced if the trough level is > 8 ng/mL. Tacrolimus will be initiated according to our practice. In this treatment arm, the Tacrolimus dose will be adjusted from day 3 on, to a target whole blood trough concentration of 4 ng/mL to 7 ng/mL. From month 2 until Month 6, the target Tacrolimus trough level will be 3 ng/mL to 6 ng/mL. After month 6, the Tacrolimus dose should be adjusted in order to achieve a target trough level of 2 ng/mL to 5 ng/mL. MMF dose will be initiated as 1 g b.i.d. (2 g/day). Adjustments should be made for adverse events including but not limited to gastrointestinal intolerance and a decrease in white blood cell (WBC).
  Other Names: Everolimus; Zortress; Tacrolimus; FK 506
  Arms: Group 2: Tacrolimus with Everolimus

SUMMARY:
The immune system is the body's defense against infection and other disease. After transplantation, the body sees the new organ as "foreign" and tries to destroy or "reject" it. Immunosuppressive medications help to prevent the immune system from attacking a transplanted organ. The primary purpose of this study is to investigate the impact of two maintenance immunosuppressive regimens. Subjects who enroll in this study will be randomly selected to have tacrolimus and everolimus (group 1) or tacrolimus and mycophenolate mofetil (group 2) as their immunosuppression medication.

This study will enroll adult patients who are scheduled to receive a kidney transplant.

The study is designed to understand the mechanisms of Everolimus in regards to kidney function in transplant recipients. The investigators hypothesis is that decreased exposure to Tacrolimus to the immune system will then translate in better renal allograft function.

DETAILED DESCRIPTION:
Immunosuppressive therapy with the calcineurin inhibitors (CNI) Cyclosporine (CsA) and Tacrolimus (Tac), have radically changed the field of organ transplantation. Ironically, although extensively and effectively used for kidney transplantation and other solid organ transplants, CsA and Tac cause important adverse renal side effects: acute and chronic renal dysfunction, hemolytic-uremic syndrome, hypertension, electrolyte disturbances and tubular acidosis. Chronic nephrotoxicity from CNI has been implicated as a principal cause of post-transplant renal dysfunction and it is characterized by an irreversible and progressive tubular atrophy, interstitial fibrosis, and focal hyalinosis of small renal arteries and arterioles. Furthermore, this class of medications is associated also, by blocking Interleukin-2 (IL2) production, with negative impact on regulatory T cells (T-Regs) generation (an important subpopulation of T helper cells that has been associated with positive immunomodulation and donor specific hypo responsiveness).

In renal transplant recipients, complete avoidance of calcineurin inhibitors from the time of renal transplant surgery has been associated with increased incidence of acute cellular rejection, and the combination of mammalian target of rapamycin (mTOR) inhibitors with full dose CNI has been shown to be synergistically nephrotoxic and it has been associated with poor graft outcome. CNI conversion to mTOR inhibitors, at different time point post-transplant, has been tested with promising results, by different investigators and by the investigators group. The investigators have shown that in a Prednisone-free immunosuppression, conversion from Tacrolimus to mTor inhibitors at different time point post transplant is safe, it is not associated with an increased risk of acute rejection and more importantly it is associated with an a persistent increase of regulatory T cells (Data presented at the American Transplant Congress (ATC) 09 and 2010) Recently the A2309 study allowed Everolimus to be FDA approved. The A2309 was a study designed to combined reduced dose Cyclosporine+Everolimus. Interesting the reduced exposure to Cyclosporine was not associated with an increase rate of albumin-creatinine ratio (ACR) and renal allograft function was well maintained compared to the control group. The A2309 opens then an important question regarding the mechanism(s) that can explain the efficacy of a low dose CNI with an mTOR inhibitor in preventing acute allograft rejection.

The present proposal is designed to understand the mechanisms of the synergistic effect(s) of low dose CNI and mTOR inhibitors (Everolimus) in controlling allo-reactive T and B cells while expanding T-Regs.

The investigators hypothesis based in published data and from their laboratory (see preliminary data-Supportive documents), is that mTOR inhibitors allow expansion of T-Regs and low exposure of CNI is sufficient to control allo-reactive T cells. Decrease exposure to CNI and concomitant increase of T-Regs will then translate in better renal allograft function and histology.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should be adults between 18 and 70 years of age
2. Subjects can be either gender or of any ethnic background
3. Subjects should be single organ recipients (kidney only)
4. Subjects must be able to understand the protocol and provide informed consent.
5. Recipient of living donor kidney transplants
6. Panel reactive antibody (PRA) < 20%

Exclusion Criteria:

1. Subjects with End Stage Renal Disease (ESRD) secondary to primary focal segmental glomerulonephritis (FSGS).
2. Inability to fully understand the purpose of the study and the inability to sign the informed consent
3. Subjects with a significant or active infection
4. Subjects who are pregnant or nursing females
5. Subjects with a history of severe hyperlipidemia not controlled with statins, patients with Cholesterol > 400mg/dl
6. Subjects with a platelet count < 100,000mm3, WBC < 2,000mm3 (or clinical practice)
7. Subjects, who, due to the existence of a surgical, medical or psychiatric condition, other than the current transplant, which in the opinion of the investigator, precludes enrollment into this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-02; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Gallon, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Donor participants were considered to be enrolled but were not part of our outcome analysis because their participation was only on the basis of providing blood for testing the immune system of the recipients.
Pre-assignment Details: Donor participants were considered to be enrolled but were not part of our outcome analysis because their participation was only on the basis of providing blood for testing the immune system of the recipients.
Period: Overall Study
Arm/Group | Group 1: Tacrolimus With MMF. | Group 2: Tacrolimus With Everolimus
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Tacrolimus With MMF. | Group 2: Tacrolimus With Everolimus | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (13) | 48.3 (16) | 48.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 20 | 20 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 11 | 18
  White | 13 | 9 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Pre-Emptive Transplant (Prior to Dialysis) [Count of Participants; unit: Participants] — Subjects that were transplanted before reaching the need to start dialysis due to end stage renal disease (ESRD).
  Participants | 7 | 6 | 13
Cause of End Stage Renal Disease [Count of Participants; unit: Participants]
  Hypertension | 5 | 6 | 11
  Polycystic Kidney Disease | 1 | 3 | 4
  Lupus | 1 | 1 | 2
  Diabetes | 10 | 5 | 15
  Unknown | 5 | 5 | 10
Induction Therapy History [Count of Participants; unit: Participants] — Type of induction therapy received by subjects prior to transplantation.
  Participants
    Alemtuzumab | 20 | 19 | 39
    IL-2 Receptor Antagonist | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in T Cell & B Cell Generation
Description: Evaluate the change in regulatory T cell generation and review the relationship of the newly generated T cells with their function in the two maintenance immunosuppressive regimens at baseline, 3 and 12 months post-transplant.
Time Frame: Baseline, 3 months, and 12 months post-transplant
Population: The percentage of Treg cells in peripheral blood is shown below per group.
Measure: Mean (Standard Deviation); unit: Mean % of Treg cells in peripheral blood
Arm/Group | Group 1: Tacrolimus With MMF. | Group 2: Tacrolimus With Everolimus
Number analyzed (Participants) | 20 | 20
Mean % of Treg cells in peripheral blood
  Baseline | 1.05 (0.17) | 0.93 (0.13)
  3 Months | 0.8 (0.19) | 1.12 (0.13)
  12 Months | 0.81 (0.10) | 1.18 (0.13)

2. Primary Outcome: Change in Glomerular Filtration Rate (GFR)
Description: Evaluate the change in graft function (as measured by GFR) at 12 months post-transplant from baseline.
Time Frame: 3 months, 6 months, and 12 months post-transplant
Measure: Mean (Standard Deviation); unit: ml/minutes per 1.73 meters^2
Arm/Group | Group 1: Tacrolimus With MMF. | Group 2: Tacrolimus With Everolimus
Number analyzed (Participants) | 19 | 20
ml/minutes per 1.73 meters^2
  3 months | 63 (19) | 66 (22)
  6 months | 64 (19) | 64 (24)
  12 months | 65 (20) | 72 (21)

3. Secondary Outcome: Patient Survival
Description: The number of patients who were alive at 2 years post transplant
Time Frame: baseline - 24 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Tacrolimus With MMF. | Group 2: Tacrolimus With Everolimus
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

4. Secondary Outcome: Renal Allograft Survival
Description: The number of subjects with renal allograft survival.
Time Frame: 12 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Tacrolimus With MMF. | Group 2: Tacrolimus With Everolimus
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

5. Secondary Outcome: Acute Rejection
Description: Number of subjects who experience acute rejection of the renal allograft.
Time Frame: 12 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Tacrolimus With MMF. | Group 2: Tacrolimus With Everolimus
Number analyzed (Participants) | 20 | 20
Participants | 4 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Group 1: Tacrolimus With MMF. | Group 2: Tacrolimus With Everolimus
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 8/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Tacrolimus With MMF. (N=20) | Group 2: Tacrolimus With Everolimus (N=20)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 3
Polyomavirus nephropathy (Infections and infestations) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Other Infection (Infections and infestations) | 3 | 5 — bacteremia, clostridium difficile colitis, abdominal abscess and herpes zoster

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT01653847/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT01653847/ICF_001.pdf